CLINICAL TRIAL: NCT03221478
Title: Effect of Kinesio Taping and Proprioceptive Exercise on the Stability of Knee in Amateur Soccer Players
Brief Title: Effect of Kinesio Taping on the Stability of Knee in Soccer Players
Acronym: KT-Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ID0018
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Injury of Musculoskeletal System
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio Taping placebo and exercises (Active Comparator): kinesio placebo and exercises
  Interventions: Other: Kinesio Taping placebo and exercises
- Kinesio Taping and exercises (Experimental): kinesio with tension and exercises
  Interventions: Other: Kinesio Taping with tension and exercises
- Kinesio Taping with tension (Experimental): Kinesio Taping with tension
  Interventions: Other: Kinesio Taping with tension

INTERVENTIONS:
Other: Kinesio Taping placebo and exercises — Kinesio Taping placebo and exercises
  Arms: Kinesio Taping placebo and exercises
Other: Kinesio Taping with tension and exercises — Kinesio Taping with tension and exercises
  Arms: Kinesio Taping and exercises
Other: Kinesio Taping with tension — Kinesio Taping with tension
  Arms: Kinesio Taping with tension

SUMMARY:
Objective: The general objective of this study is to determine the possible beneficial effect of the application of kinesiotaping, as well as the performance of proprioceptive exercises on parameters related to knee stability, such as the incidence of injuries, pain, static stability Or dynamics, and flexibility, in amateur soccer players, with a workload of 3 days per week plus the match.

Material and methods: Amateur soccer players are divided into 3 groups.

Group 1 (G1) performs proprioceptive exercises plus the application of kinesiotaping without tension in the knee.

Group 2 (G2) performs proprioceptive exercises plus the application of kinesiotaping with tension in the knee.

Group 3 (G3) is placed kinesiotaping with tension in the knee, without proprioception exercises.

The treatment will last four weeks and three evaluations, one before treatment, another at two weeks and the last one at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Football players
* Over 18 years with experience in this sport over 5 years

Exclusion Criteria:

* Players with pathologies that prevented them from playing football normally
* Recent serious injuries
* Allergy to kinesiotaping
* Impossibility to complete the study

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 46 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
KOOS knee questionnaire | 4 weeks

SECONDARY OUTCOMES:
Star Excursion Balance Test (SEBT) | 4 weeks
Unipedal Stance Test (UST) | 4 weeks
Sit and reach (Toe touch test) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gemma V Espí-López, Principal Investigator — University of Physiotherapy
Locations (1):
- Gemma Victoria Espí-López, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No